CLINICAL TRIAL: NCT07302659
Title: Surgical Techniques to Prevent Perioperative Neurologic Complications in Patients Undergoing Coronary Artery Bypass Grafting
Acronym: PROTECT-CABG
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2023ZD0504701
Record Dates: First submitted 2025-11-19; First posted 2025-12-24 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Coronary Artery Bypass Graft (CABG)
Keywords: coronary artery bypass graft; Silent Brain Infarction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional off-pump coronary artery bypass grafting (AO-SVG) (No Intervention)
- Aortic no-touch coronary artery bypass grafting (RIMA-SVG) (Experimental)
  Interventions: Procedure: Aortic no-touch coronary artery bypass grafting (RIMA-SVG)

INTERVENTIONS:
Procedure: Aortic no-touch coronary artery bypass grafting (RIMA-SVG) — Ascending aortic no-touch CABG with saphenous vein graft (SVG) anastomosed to the right internal mammary artery (RIMA)
  Arms: Aortic no-touch coronary artery bypass grafting (RIMA-SVG)

SUMMARY:
To explore surgical strategies that reduce perioperative neurologic complications in cardiovascular surgery, with the aim of improving perioperative outcomes and quality of life while reducing the socioeconomic burden. Specifically:

This multicenter, randomized controlled clinical trial will evaluate the benefits of a novel aortic no-touch technique in reducing perioperative silent brain infarction(SBI) among patients undergoing surgical treatment for coronary artery disease. The findings are expected to provide a safe and effective myocardial revascularization strategy for individuals at high risk of cerebral ischemia.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>18 years old) with multivessel coronary artery disease who are scheduled to undergo isolated off-pump coronary artery bypass grafting and who provide informed consent to participate in this study.

Exclusion Criteria:

* Indications for cardiopulmonary bypass surgery (or no contraindications to on-pump surgery);
* Great saphenous vein is unsuitable for use as a graft conduit;
* Subclavian artery stenosis or occlusion, or any contraindication to the use of the internal mammary artery as a graft conduit;
* History of previous cardiac surgery;
* Emergency surgery;
* Inability to apply an aortic clamp due to severe ascending aortic calcification;
* Expected inability to tolerate MRI or contraindications to MRI (e.g., known intolerance to MRI, an implanted permanent pacemaker, or an anticipated need for permanent pacemaker implantation);
* Inability to complete neurocognitive assessment due to language barriers or visual/hearing impairment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Estimated)
Dates: Start 2026-02-14 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Saphenous vein graft (SVG) occlusion rate | 1 year after surgery
  Assessed by coronary computed tomography angiography (CCTA)
New-onset clinical stroke and silent brain infarction (SBI) | 7 ± 3 days after surgery
  Clinical stroke and SBI assessed at 7 ± 3 days postoperatively; SBI assessed by brain magnetic resonance imaging (MRI).

SECONDARY OUTCOMES:
Incidence of postoperative delirium | within 5 postoperative days
  The incidence of delirium evaluated by CAM/CAM-ICU
Incidence of perioperative neurocognitive disorder (PND) | within 7 days after surgery
  Cognitive function will be assessed using the Montreal Cognitive Assessment (MoCA)
Perioperative major adverse cardiovascular and cerebrovascular events (MACCE) | within 30 postoperative days
  Major adverse cardiovascular and cerebrovascular events are defined as the composite of all-cause death, myocardial infarction, stroke and repeat revascularization.
MACCE within 3 months after surgery | Up to 3 months after surgery (3-month follow-up)
  Major adverse cardiovascular and cerebrovascular events are defined as the composite of all-cause death, myocardial infarction, stroke and repeat revascularization.
Clinical stroke within 3 months after surgery | Up to 3 months after surgery (3-month follow-up)
Sternal complications within 3 months after surgery | Up to 3 months after surgery (3-month follow-up)
Cognitive dysfunction at 3 months after surgery | 3 months after surgery
  Cognitive function will be assessed using the Montreal Cognitive Assessment (MoCA).
Angina within 12 months after surgery | 12 months after surgery
  Patients will complete the Seattle Angina Questionnaire (SAQ) at baseline pre-procedure and again at 12 months post CABG
Cognitive dysfunction at 12 months after surgery | 12 months after surgery
  Cognitive function will be assessed using the Montreal Cognitive Assessment (MoCA).
Sternal complications within 12 months after surgery | Up to 12 months after surgery (12-month follow-up)
Clinical stroke within 12 months after surgery | Up to 12 months after surgery (12-month follow-up)
MACCE within 12 months after surgery | Up to 12 months after surgery (12-month follow-up)
  Major adverse cardiovascular and cerebrovascular events are defined as the composite of all-cause death, myocardial infarction, stroke and repeat revascularization.

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Fuwai Hospital Chinese Academy of Medical Sciences, Beijing
  - Peking University First Hospita, Beijing
  - Qingdao Cardiovascular Hospital, Qingdao
  - Fuwai Hospital Chinese Academy of Medical Sciences, Shenzhen, Shenzhen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zhao DF, Edelman JJ, Seco M, Bannon PG, Wilson MK, Byrom MJ, Thourani V, Lamy A, Taggart DP, Puskas JD, Vallely MP. Coronary Artery Bypass Grafting With and Without Manipulation of the Ascending Aorta: A Network Meta-Analysis. J Am Coll Cardiol. 2017 Feb 28;69(8):924-936. doi: 10.1016/j.jacc.2016.11.071. PMID 28231944
- [Result] Tachibana H, Hiraoka A, Saito K, Naito Y, Chikazawa G, Tamura K, Totsugawa T, Yoshitaka H, Sakaguchi T. Incidence and impact of silent brain lesions after coronary artery bypass grafting. J Thorac Cardiovasc Surg. 2021 Feb;161(2):636-644. doi: 10.1016/j.jtcvs.2019.09.162. Epub 2019 Oct 16. PMID 31735394